CLINICAL TRIAL: NCT05703412
Title: Effectiveness of a Multi-component mHealth Intervention to Improve Post-hospital Transitions of Care for Patients With SMI
Brief Title: Effectiveness of mHealth Post-discharge Intervention for Patients With Severe Mental Illness
Acronym: tFOCUS
Status: Enrolling by invitation | Phase: Not Applicable | Type: Interventional
Sponsor: Butler Hospital (Other)
Collaborators: National Institute of Mental Health (NIMH) (NIH); Brown University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 2208-001; R01MH130496 (NIH)
Record Dates: First submitted 2023-01-19; First posted 2023-01-30 (Actual); Last update posted 2025-06-06 (Actual); Status verified 2025-06

CONDITIONS: Bipolar Disorder; Major Depression; Schizophrenia
Keywords: mHealth; psychiatric hospitalization; transitions of care
MeSH Terms: conditions — Bipolar Disorder; Depressive Disorder, Major; Schizophrenia

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Transition-FOCUS mHealth Intervention (Experimental): All participants will download the tFOCUS app to their mobile phone. tFOCUS uses EMA to assess variables identified as being salient to treatment engagement and illness self-management. The application delivers algorithm-driven micro interventions to address reported problem(s). Data is transmitted to a clinician "dashboard," which can be used for remote monitoring.
  Interventions: Behavioral: Transition-FOCUS mHealth Intervention
- Check-In (Active Comparator): Control participants will receive the currently recommended best practices of post-discharge care, including follow-up appointments, instructions, referrals and a follow-up check in.
  Interventions: Behavioral: Check-In

INTERVENTIONS:
Behavioral: Transition-FOCUS mHealth Intervention — tFOCUS integrates evidence-based strategies for self-management of severe mental illness (SMI) into a comprehensive mobile assessment and treatment system that is grounded in theoretical SMI models. The application promotes self-management strategies aimed at improving medication adherence to manage biologically driven psychiatric symptoms, increase social support to reduce the negative impact of social withdrawal, improve sleep hygiene to reduce levels of fatigue, and promote strategies for coping with persistent symptoms. tFOCUS application strategies are linked to participants' specific assessment responses, allowing for a highly personalized self-management intervention experience
  Other Names: tFOCUS
  Arms: Transition-FOCUS mHealth Intervention
Behavioral: Check-In — Check-in includes a discharge and safety plan (with medication instructions, crisis services, etc.), a timely follow-up appointment with a mental health provider, and phone check-ins by case managers immediately following post-discharge for care coordination purposes.
  Arms: Check-In

SUMMARY:
The overall aim of this program of research is to improve the continuity of care for patients with serious mental illness (SMI) by supporting a safer and more efficient bridge from hospital to outpatient care using a mobile device-delivered app called Transition-FOCUS (tFOCUS), which has previously been tested in community samples. The purpose of the proposed project is to establish the effectiveness of our empirically-supported, multi-component mHealth intervention.

ELIGIBILITY:
Inclusion Criteria:

* psychiatric inpatient/partial hospitalization
* diagnosis of schizophrenia-spectrum disorder or major mood disorder
* planned ongoing mental health treatment post-discharge in the community
* 18 years or older
* ability to speak and read English

Exclusion Criteria:

* lack of smartphone
* homelessness or housing instability that would prevent reliable follow-up
* discharge to a long-term restricted living setting

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 180 (Estimated)
Dates: Start 2023-02-14 (Actual); Primary Completion 2027-07-31 (Estimated); Study Completion 2027-07-31 (Estimated)

PRIMARY OUTCOMES:
Brief Psychiatric Rating Scale (BPRS) | 24 weeks
  The interviewer-rated Brief Psychiatric Rating Scale is a measure of psychiatric symptom severity. The total score (sum of items) will be used to assess overall severity with scores ranging from 18 to 126 and higher scores indicating greater severity.

OTHER OUTCOMES:
Recovery Assessment Scale (RAS) | 24 weeks
  The RAS is a self-report measure of aspects of mental health recovery, including hope and self-determination. The total score (sum of items) will be used and ranges from 22 to 110 with higher scores indicating higher suicidal thoughts and behaviors.

CONTACTS AND LOCATIONS:
Overall Officials: Brandon Gaudiano, PhD, Principal Investigator — Butler Hospital; Ethan Moitra, PhD, Principal Investigator — Brown University
Locations (1):
- Butler Hospital, Providence, Rhode Island, United States

IPD SHARING:
Plan to Share IPD: Yes
Data will be uploaded to the NIMH Data Archive.
Supporting Information: Study Protocol
Time Frame: De-identified data will be available after the project is completed without time limit.
Access Criteria: See guidelines of the NIMH Data Archive.
URL: https://nda.nih.gov/

REFERENCES:
- [Derived] Moitra E, Amaral TM, Benz MB, Cambow S, Elwy AR, Kunicki ZJ, Lu Z, Rafferty NS, Rabasco A, Rossi R, Schatten HT, Gaudiano BA. A Hybrid Type 1 trial of a multi-component mHealth intervention to improve post-hospital transitions of care for patients with serious mental illness: Study protocol. Contemp Clin Trials. 2024 Apr;139:107481. doi: 10.1016/j.cct.2024.107481. Epub 2024 Mar 1. PMID 38431134